CLINICAL TRIAL: NCT02149719
Title: Phase 2 Randomised Study of Oral Immunotherapy Using Boiled Peanut to Induce Desensitisation in Children With Challenge-proven, IgE-mediated Peanut Allergy
Brief Title: Boiled Peanut Oral Immunotherapy for the Treatment of Peanut Allergy: a Pilot Study
Acronym: BOPI-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Sydney (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Paul Turner, Principal Investigator, Imperial College London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15SM2492; ACTRN12614000265673 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2014-05-24; First posted 2014-05-29 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: IgE Mediated Peanut Allergy
Keywords: Peanut allergy; Desensitisation; Safety
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desensitisation to peanut (Experimental): Desensitisation using boiled peanut
  Interventions: Other: Desensitisation using boiled peanut
- Control (Experimental): Subjects allocated to the control group will undergo routine care for 12 months, following which they will be offered the active treatment with boiled peanut (as a one-way cross-over intervention).
  Interventions: Other: Desensitisation using boiled peanut (deferred start)

INTERVENTIONS:
Other: Desensitisation using boiled peanut
  Arms: Desensitisation to peanut
Other: Desensitisation using boiled peanut (deferred start)
  Arms: Control

SUMMARY:
Peanut allergy is increasingly common, especially in countries such as UK and Australia. There is currently no accepted routine clinical therapy to cure peanut allergy. Recently studies have looked at desensitising people with peanut allergy by giving them small daily doses of roasted peanut. Although this therapy works for some people, its effects are not generally long lasting and it is associated with many side effects during protocol, resulting in a significant rate of drop-outs.

Pilot data suggests that boiled peanut is less immunogenic than roasted peanut, and may therefore provide a safer way of inducing desensitisation in patients who are allergic to roasted peanut, by first inducing tolerance to boiled peanut.

Study hypothesis: Increasing doses of boiled peanut can induce desensitisation to roasted peanut, in peanut-allergic individuals.

ELIGIBILITY:
Inclusion Criteria:

* IgE-mediated peanut allergy, confirmed at double-blind placebo-controlled food challenge
* Tolerant to at least 1/4 boiled peanut (boiled for 4 hours) at open food challenge.
* Informed consent of parent/legal guardian and patient assent

Exclusion Criteria:

* Allergic to 1/4 boiled peanut at PCFC
* Tolerates ≥1.4 g roasted peanut protein at entry PCFC
* Unstable asthma
* Unwilling or unable to fulfil study requirements
* Undergoing other forms of immunotherapy (e.g. SCIT or SLIT to aeroallergens)
* Previous admission to ICU for management of allergic reaction to peanut
* Clinically significant chronic illness (other than asthma, rhinitis or eczema).
* Undergoing subcutaneous or sublingual immunotherapy and within the first year of therapy, for respiratory allergy.
* Subjects receiving anti-IgE therapy, oral immunosupressants, beta-blocker or ACE inhibitor therapy.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dianne E Campbell, FRACP PhD, Study Chair — The Children's Hospital at Westmead, Australia; Sam Mehr, FRACP, Study Director — The Children's Hospital at Westmead, Australia; Paul J Turner, FRACP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London / Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Turner PJ, Ruiz-Garcia M, Patel N, Abrantes G, Burrell S, Vazquez-Ortiz M, Skypala I, Durham SR, Boyle RJ. Delayed symptoms and orthostatic intolerance following peanut challenge. Clin Exp Allergy. 2021 May;51(5):696-702. doi: 10.1111/cea.13865. Epub 2021 Mar 21. PMID 33715235
- [Derived] Burrell S, Patel N, Vazquez-Ortiz M, Campbell DE, DunnGalvin A, Turner PJ. Self-administration of adrenaline for anaphylaxis during in-hospital food challenges improves health-related quality of life. Arch Dis Child. 2021 Jun;106(6):558-563. doi: 10.1136/archdischild-2020-319906. Epub 2020 Sep 18. PMID 32948514

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Subjects allocated to the control group will undergo routine care for 12 months, following which they will be offered the active treatment with boiled peanut (as a one-way cross-over intervention).
  Desensitisation using boiled peanut (deferred start)
Period: Overall Study
Arm/Group | Desensitisation to Peanut | Control
Started | 32 | 15
Completed | 24 | 14
Not Completed | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desensitisation to Peanut | Control | Total
Number analyzed (Participants) | 32 | 15 | 47
Age, Continuous [Median (Full Range); unit: years] | 12.5 [8 to 16.9] | 12.5 [8.9 to 15.4] | 12.5 [8 to 16.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 21 | 6 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 32 | 15 | 47
Diagnosis of asthma [Count of Participants; unit: Participants] | 20 | 12 | 32
Previous anaphylaxis to peanut [Count of Participants; unit: Participants] | 14 | 5 | 19
Skin prick test to commercial peanut allergen [Median (Full Range); unit: mm skin wheal] | 9 [3 to 22] | 9 [6 to 17] | 9 [3 to 22]
Serum IgE to peanut [Median (Full Range); unit: kUA/lL] | 32.9 [0.9 to 412] | 38.7 [1.2 to 247] | 35.8 [0.9 to 412]
Serum IgE to ara h 2 [Median (Full Range); unit: kUA/lL] | 17 [0.5 to 248] | 32.8 [0.8 to 173] | 17.4 [0.5 to 248]

OUTCOME MEASURES:

1. Primary Outcome: Desensitisation to >1.4g (Roasted) Peanut Protein at Food Challenge
Description: The proportion of participants who tolerate 1.4g (or more) roasted peanut protein after 12 months of OIT as assessed by DBPCFC, in the active vs control group.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Desensitisation to Peanut | Control
Number analyzed (Participants) | 32 | 15
Participants | 24 | 14
Statistical Analysis 1: Comparison: Desensitisation to Peanut vs Control; Test type: Superiority; p < 0.0001, Fisher Exact

2. Secondary Outcome: Change in Threshold to Roasted Peanut After 6 and 12 Months of OIT
Description: Relative change in clinical threshold (No observed adverse event level, NOAEL; Lowest observed adverse event level, LOAEL) to roasted peanut at 6 and 12 months.
Time Frame: 6 and 12 months after study intervention
Reporting Status: Not Posted

3. Secondary Outcome: Sustained Unresponsiveness After 4 Week Cessation of Maintenance OIT
Description: Rate of sustained unresponsiveness after 4 week cessation of maintenance OIT at 1 year.
Time Frame: After 1 year of OIT
Reporting Status: Not Posted

4. Secondary Outcome: Safety, Incidence of Adverse Event
Description: Incidence of adverse allergic events during desensitisation protocol
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life Measures
Description: Quality of Life assessment and how this changes during peanut desensitisation.
Time Frame: 6, 12 and 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Study Compliance
Description: Compliance with study protocol
Time Frame: 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Immunological Outcomes
Description: Immunological outcome measures pre-, during and post- 12 months of OIT
Time Frame: Pre, 3, 6, and 12 months post start of OIT
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Threshold in Peanut-allergic Subjects Found to be Tolerant to Boiled Peanut at Baseline
Description: Change in threshold in peanut-allergic subjects found to be tolerant to boiled peanut at baseline, as determined by double-blind, placebo-controlled food challenges pre- and post- desensitisation.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year (2 years in control arm)
Groups:
- Control - Avoidance Phase: Subjects allocated to the control group will undergo routine care for 12 months, following which they will be offered the active treatment with boiled peanut (as a one-way cross-over intervention).
- Control - Desensitisation Phase: Subjects allocated to the control group underwent routine care (dietary avoidance) for 12 months, following which they were offered active treatment with boiled peanut (as a one-way cross-over intervention).
Arm/Group | Desensitisation to Peanut | Control - Avoidance Phase | Control - Desensitisation Phase
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 17/32 | 6/15 | 3/15
Other Adverse Events (participants affected / at risk) | 32/32 | 0/15 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desensitisation to Peanut (N=32) | Control - Avoidance Phase (N=15) | Control - Desensitisation Phase (N=15)
Uncomplicated anaphylaxis at hospital food challenge (Immune system disorders) | 12 (25) | 6 (10) | 0 (0)
Anaphylaxis due to dosing at home (Immune system disorders) | 11 (21) | 0 (0) | 3 (4)
Anaphylaxis not related to study intervention (Immune system disorders) | 1 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desensitisation to Peanut (N=32) | Control - Avoidance Phase (N=15) | Control - Desensitisation Phase (N=15)
Allergic reaction due to study intervention (Immune system disorders) | 32 (1017) | 0 (0) | 12 (115) — In year 1 of study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02149719/Prot_SAP_000.pdf